CLINICAL TRIAL: NCT06057194
Title: Prospective Study to Assess the Efficacy of Letermovir Prophylaxis in Preventing CMV Infection in Lung Transplant Recipients Compared to a Retrospective Cohort Treated With Standard Valganciclovir Prophylaxis for 12 Months (LETERCOR Study)
Brief Title: Efficacy of Letermovir in Preventing Cytomegalovirus (CMV) Infection in Lung Transplant Recipients vs. Valganciclovir.
Acronym: LETERCOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: MERCK SHARP & DOHME DE ESPAÑA S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCO-LET-2022-01; 2023-504384-16-00 (Other: EMA)
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Infections, Cytomegalovirus
Keywords: Lung transplant; CMV prophylaxis; Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir; Tablets

STUDY DESIGN:
Intervention Model Description: Clinical trial of a prospective cohort compared to a retrospective (historical control) cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letermovir (prospective cohort) (Experimental): 2 tablets of 240 milligrams (mg) Letermovir orally once daily. during 12 months
  Interventions: Drug: Letermovir 240 mg Oral Tablet
- Valganciclovir (retrospective cohort) (No Intervention): Retrospective cohort, of patients treated with Valganciclovir during 12 months

INTERVENTIONS:
Drug: Letermovir 240 mg Oral Tablet — Treatment will commence as soon as subjects can receive oral medication, with a maximum timeframe of 28 days after transplantation. If patients cannot receive oral medication after transplantation, initial prophylaxis with ganciclovir per clinical practice will be allowed. Medication will be discontinued 12 months after treatment initiation.
  Arms: Letermovir (prospective cohort)

SUMMARY:
The goal of this quasi-experimental multicenter before-after cohort study, phase II study is to evaluate the efficacy of 12-month letermovir prophylaxis in lung transplant recipients (D+/R-) compared to a historical cohort of lung transplant recipients (D+/R-) who received 12 months of valganciclovir prophylaxis to prevent CMV disease."

ELIGIBILITY:
Inclusion Criteria (prospective cohort):

* Adults over 18 years old
* Lung transplant recipients (D+/R-) pre-transplant.
* Having an undetectable CMV polymerase chain reaction assay (PCR) within the 96 hours prior to the start of letermovir prophylaxis.
* Patients who have provided written informed consent.

Exclusion Criteria (prospective cohort):

* HIV-infected patients.
* Patients with multivisceral transplant.
* Patients unable to comply with the follow-up protocol.
* Receiving a different antiviral prophylaxis other than ganciclovir prior to letermovir prophylaxis.
* Patients with concurrent renal and hepatic insufficiency.

Inclusion Criteria (retrospective cohort):

* Adults over 18 years old. Lung transplant recipients (D+/R-) pre-transplant.
* Patients treated with Valganciclovir prophylaxis for 12 months.
* Patients transplanted within 2 years prior to the start of the study.
* Patients with a complete 13-month follow-up and comparable data to the prospective cohort to evaluate the study's primary variables.

Exclusion Criteria (retrospective cohort):

* HIV-infected patients.
* Patients with multivisceral transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV disease/replication | During 12 months after initiation of prophylaxis
  CMV replication: The term 'replication' can be used to indicate evidence of multiplication and is sometimes used interchangeably with CMV infection
  CMV disease: It is defined as symptomatic replication or invasive disease of organs or tissues that requires treatment at the investigator's discretion."

SECONDARY OUTCOMES:
Antiviral prophylaxis received: | During 12 months after initiation of prophylaxis
  Doses administered of Letermovir or Valganciclovir
Dose of non anti-viral CMV Medications: Any non-antiviral therapy received as standard of care (SoC) for the management of CMV (e.g., immunoglobulins) | During 12 months after initiation of prophylaxis
  Drug Dose (mg/hour)
Administration route of non-antiviral CMV Medications: Any non-antiviral therapy received as standard of care (SoC) for the management of CMV (e.g., immunoglobulins) | During 12 months after initiation of prophylaxis
  Drug Administration Route
Duration of treatment of non-antiviral CMV Medications: Any non-antiviral therapy received as standard of care (SoC) for the management of CMV (e.g., immunoglobulins) | During 12 months after initiation of prophylaxis
  Drug treatment duration (days)
Discontinuation of non-antiviral CMV Medications: Any non-antiviral therapy received as standard of care (SoC) for the management of CMV (e.g., immunoglobulins) | During 12 months after initiation of prophylaxis
  Drug Reason for Discontinuation
Reduction of the antiviral dose related to CMV antiviral toxicity | During 12 months after initiation of prophylaxis
  Number of events of reduction
Substitution of letermovir by intravenous ganciclovir or foscarnet IV, related to CMV antiviral toxicity | During 12 months after initiation of prophylaxis
  Number of substitutions
Dose changes of immunosuppressive therapy related to CMV antiviral toxicity | During 12 months after initiation of prophylaxis
  Number of changes
Changes of immunosuppressive therapy related to CMV antiviral toxicity | During 12 months after initiation of prophylaxis
  Number of changes
Use of granulocyte colony-stimulating factors (G-CSF). | During 12 months after initiation of prophylaxis
  Number of events (use)
Incidence of leucopenia | During 12 months after initiation of prophylaxis
  Incidence of leucopenia. (leucopenia will be considered if the total leukocyte count is less than 3,000/mL)
Incidence of neutropenia | During 12 months after initiation of prophylaxis
  Incidence of leucopenia. (neutropenia will be considered if the total neutrophil count is less than 1,000/mL)
Hospital readmission associated with CMV complication | During 12 months after initiation of prophylaxis
  Number of events
Incidence of viral, bacterial, or opportunistic fungal infections during the study follow-up period. | During 12 months after initiation of prophylaxis
  Number of events
Incidence of renal toxicity directly related to CMV antivirals. | During 12 months after initiation of prophylaxis
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Julián C De la Torre Cisneros, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Córdoba, Spain